CLINICAL TRIAL: NCT01610310
Title: A Randomized, Open-Label, Crossover Phase 1 Study to Evaluate the Pharmacokinetic Profile, Safety, and Tolerability of Peginterferon Beta-1a (BIIB017) Delivered by Pre-filled Syringe (PFS) or Autoinjector in Healthy Volunteers
Brief Title: Peginterferon Beta-1a (BIIB017) Autoinjector Pharmacokinetic Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 105HV103
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Healthy; Multiple Sclerosis
Keywords: SC; PEG; Inteferon; PK; Subcutaneous; PEGylated; Autoinjector; Injectable; MS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- peginterferon beta-1a PFS/autoinjector (Experimental): A single dose of peginterferon beta-1a 125 mcg administered by prefilled syringe (PFS) on Day 1, then by a single dose of peginterferon beta-1a 125 mcg by autoinjector on Day 22.
  Interventions: Device: BIIB017 (peginterferon beta-1a) Pre-filled syringe (PFS); Device: BIIB017 (peginterferon beta-1a) Autoinjector
- peginterferon beta-1a autoinjector / PFS (Experimental): A single dose of peginterferon beta-1a 125 mcg administered by autoinjector on Day 1, then by a single dose of peginterferon beta-1a 125 mcg by prefilled syringe (PFS) on Day 22.
  Interventions: Device: BIIB017 (peginterferon beta-1a) Pre-filled syringe (PFS); Device: BIIB017 (peginterferon beta-1a) Autoinjector

INTERVENTIONS:
Device: BIIB017 (peginterferon beta-1a) Pre-filled syringe (PFS) — 125 mcg of peginterferon beta-1a (BIIB017) subcutaneous injection (SC) administered by PFS once on either Day 1 or Day 22
  Other Names: BIIB017
Device: BIIB017 (peginterferon beta-1a) Autoinjector — 125 mcg of peginterferon beta-1a (BIIB017) subcutaneous injection (SC) administered by autoinjector once on either Day 1 or Day 22
  Other Names: BIIB017

SUMMARY:
The purpose of this study is to characterize the pharmacokinetic (PK) profile, safety, and tolerability of peginterferon beta-1a (BIIB017) delivered by the single-use autoinjector or prefilled syringe (PFS) in healthy volunteers to support the development of the autoinjector.

DETAILED DESCRIPTION:
This is a randomized, open-label, 2-sequence, 2-period crossover study that will be conducted at a single site in the United States to characterize the PK profile, safety and tolerability of peginterferon beta-1a delivered by autoinjector or PFS. Participants will be randomized in a 1:1 ratio to receive a single dose of peginterferon beta-1a at Day 1 delivered by either autoinjector or PFS, followed by a single dose of peginterferon beta 1a delivered by the other device at Day 22. The total duration of study participation is up to 3 months for each participant. Participants will complete a follow-up visit at Day 50 after the end of treatment period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Must have a body mass index (BMI) of 19 to 29 kg/m^2, inclusive, and a minimum body weight of 50.0 kg

Key Exclusion Criteria:

1. History of any clinically significant laboratory abnormalities, malignancies, cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major diseases
2. Female subjects who are pregnant or breastfeeding
3. Any previous treatment with prescription or investigational pegylated drugs.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Area under the time-concentration curve for serum concentrations of peginterferon beta-1a from time zero to infinity post dose (AUC0-∞) | For 11 days (multiple timepoints) after each dose on Day 1 and 22

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of peginterferon beta-1a | For 11 days (multiple timepoints) after each dose on Day 1 and 22
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 up to Day 50
Changes in clinical laboratory assessments | Day 1 up to Day 50
Vital sign changes | Day 1 up to Day 50)
Physical exam changes | Day 1 up to Day 50
Electrocardiogram changes | Day 1 up to Day 50
Clinician injection site assessment | Days 1+2, 22+23

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Saint Paul, Minnesota, United States